CLINICAL TRIAL: NCT00586209
Title: A Phase II, Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Study of L Glutamine Therapy for Sickle Cell Anemia and Sickle ß0-Thalassemia
Brief Title: L-Glutamine Therapy for Sickle Cell Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate clinical supplies and Emmaus business decision.
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Emmaus Medical, Inc. (Industry)
Responsible Party: Principal Investigator, yutaka niihara, President, Emmaus Medical, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10511-01RY
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Sickle Cell Anemia; Thalassemia
Keywords: sickle cell disease; sickle cell anemia; L-glutamine; Sickle Cell Anemia (homozygous); Sickle β°-Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-glutamine (Experimental): L-glutamine group will be given at the following dosage:
  17-33.3 kg at 5 g 2x daily 33.4-66.6 kg at 10 g 2X daily >66.7 at 15 g 2X daily
  Interventions: Drug: L-Glutamine
- Placebo (Placebo Comparator): Maltodextrin group will be given at the following dosage:
  17-33.3 kg at 5 g 2x daily 33.4-66.6 kg at 10 g 2X daily >66.7 at 15 g 2X daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-Glutamine — L-Glutamine at: 5 g 2X daily (17-33.3 Kg) 10 g 2x daily (33.4-66.6 Kg) 15 g 2x daily (>66.7 kg)
  Arms: L-glutamine
Drug: Placebo — Placebo (75% Maltodextrin, 24.5 % Starch, 0.5% Tricalcium Phosphate) - given at the same dosage as L-glutamine
  Arms: Placebo

SUMMARY:
The primary purpose is to evaluate the effect of L-glutamine therapy on exercise endurance and breath by breath exercise response of sickle cell anemia patients

The secondary purpose is to assess the effect of L-glutamine on incidence of painful crises; level of chronic pain, and amount of daily requirement for narcotics.

DETAILED DESCRIPTION:
This is a phase II, prospective, randomized, double-blind, placebo-controlled, parallel-group,study to evaluate the safety and efficacy of oral L-glutamine therapy for patients with sickle cell anemia or sickle β°-thalassemia who are at least 18 years old with focus on the aspect of exercise endurance. In this study, the patients will orally take L-glutamine or placebo twice daily, and clinical and hematological parameters will be monitored. The adverse events,especially those attributable to L-glutamine therapy, will also be monitored.

The data obtained will be essential in understanding the role of L-glutamine in therapy for sickle cell anemia and sickle β°-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the study, a patient must meet all of the following inclusion criteria:

* Patient is at least 18 years of age.
* Patient has been diagnosed with sickle cell anemia or sickle ß0-thalassemia (documented by hemoglobin electrophoresis).
* Patient has had at least two episodes of painful crises within 12 months of the screening visit.
* If the patient has been treated with an anti-sickling agent within three months of the screening visit, the therapy must have been continuous for at least three months with the intent to continue for the next 14 months.
* Patient or the patient's legally authorized representative has given written informed consent.
* If the patient is a female of child-bearing potential, she agrees to practice a recognized form of birth control during the course of the study.
* Patient is able to perform exercise tolerance test

Exclusion Criteria:

If the patient meets any of the following criteria, the patient must not be enrolled:

* Patient has a significant medical condition that required hospitalization (other than sickle painful crisis) within two months of the screening visit.
* Patient has diabetes mellitus with untreated fasting blood sugar >115 mg/dL.
* Patient has prothrombin time International Normalized Ratio (INR) > 2.0.
* Patient has serum albumin < 3.0 g/dl.
* Patient has received any blood products within three weeks of the screening visit.
* Patient has a history of uncontrolled liver disease or renal insufficiency.
* Patient is pregnant or lactating.
* Patient has been treated with an experimental anti-sickling medication/treatment (except hydroxyurea) within 30 days of the screening visit.
* Patient has been treated with an experimental drug within 30 days of the screening visit.
* There are factors that would, in the judgment of the investigator, make it difficult for the patient to comply with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-02-06 (Actual); Primary Completion 2008-08-27 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Niihara, MD, Principal Investigator — LaBiomed At Harbor-UCLA Medical Center
Locations (1):
- LA Biomed at Harbor-UCLA Medical Center, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- L-glutamine: L-glutamine group will be given at the following dosage:
  17-33.3 kg at 5 g 2x daily 33.4-66.6 kg at 10 g 2X daily >66.7 at 15 g 2X daily
  L-Glutamine: L-Glutamine at: 5 g 2X daily (17-33.3 Kg) 10 g 2x daily (33.4-66.6 Kg) 15 g 2x daily (>66.7 kg)
- Placebo: Maltodextrin group will be given at the following dosage:
  17-33.3 kg at 5 g 2x daily 33.4-66.6 kg at 10 g 2X daily >66.7 at 15 g 2X daily
  Placebo: Placebo (75% Maltodextrin, 24.5 % Starch, 0.5% Tricalcium Phosphate) - given at the same dosage as L-glutamine
Period: Overall Study
Arm/Group | L-glutamine | Placebo
Started | 5 | 10
Completed | 5 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-glutamine | Placebo | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Effect of L-glutamine Therapy on Exercise Endurance of Sickle Cell Anemia Patients
Description: Exercise endurance will be examined at each visit. Change from baseline will be reported at weeks 8 and 12
Time Frame: Baseline, Weeks 8 and 12
Population: The study was terminated by the Sponsor's business decision prior to achieving the planned enrollment. Due to this the data was not collected and not analyzed. However safety data was collected and analyzed to gather data on the safety of L-glutamine in sickle cell patients.
Arm/Group | L-glutamine | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Effect of L-glutamine Therapy on Breath by Breath Exercise of Sickle Cell Patients
Description: Breath by breath exercise will be examined at each visit. Change from baseline will be reported at weeks 8 and 12
Time Frame: Baseline, Weeks 18 and 12
Population: as for outcome 1
Arm/Group | L-glutamine | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Effect of Oral L-glutamine on Incidence of Painful Crises
Description: Incidence of panful crises will be assessed at each visit.
Time Frame: From Week 0 through Week 12
Population: as for outcome 1
Arm/Group | L-glutamine | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Effect of Oral L-glutamine on Amount of Daily Requirement for Narcotics
Description: Amount of daily requirement for narcotics will assessed at each visit.
Time Frame: From Week 0 through Week 20
Population: as for outcome 1
Arm/Group | L-glutamine | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Effect of Oral L-glutamine on Level of Chronic Pain
Description: Level of chronic pain will be assessed at each visit.
Time Frame: From Week 0 to Week 12
Population: as for outcome 1
Arm/Group | L-glutamine | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected throughout the course of the study (53 weeks or about 1 year).
Description: The Safety population will include all patients who received at least one dose of study medication.
Arm/Group | L-glutamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/5 | 5/10
Other Adverse Events (participants affected / at risk) | 4/5 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-glutamine (N=5) | Placebo (N=10)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 (1) | 4 (4)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-glutamine (N=5) | Placebo (N=10)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No